CLINICAL TRIAL: NCT04218045
Title: Laparoscopic Single Anastomosis Sleeve Ileal (SASI) Bypass Versus Laparoscopic Sleeve Gastrectomy For Morbidly Obese Patients
Brief Title: Laparoscopic Single Anastomosis Sleeve Ileal Bypass Versus Laparoscopic Sleeve Gastrectomy For Morbidly Obese Patients
Acronym: SASI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, yousef ahmed el-ayman, assistant lecturer of general surgery, Master degree, MD Candidate, Zagazig University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YousefMDThesis
Record Dates: First submitted 2019-01-08; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Bariatric Surgery
Keywords: sleeve; laparoscopy; SASI; Morbid obesity; metabolic surgery; gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Non-randomized controlled trial, where patients are assigned to one of two kinds of bariatric procedures, and results are compared between both groups
Masking Description: Masking cannot be applied as both patient and surgeons must be fully informed and consenting regarding the procedure of choice, and the possible outcomes and complications
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic sleeve gastrectomy group (Active Comparator): The group of morbidly obese patients undergoing laparoscopic sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- SASI bypass group (Experimental): The group of morbidly obese patients undergoing laparoscopic single- anastomosis sleeve ileal bypass (the new procedure being evaluated)
  Interventions: Procedure: Laparoscopic single anastomosis sleeve ileal bypass

INTERVENTIONS:
Procedure: Laparoscopic single anastomosis sleeve ileal bypass — a simple loop gastro-ileal bypass is added to the sleeve procedure.
  Other Names: SASI bypass - Santoro's operation - sleeve gastrectomy with transit bipartite - SG þ TB
  Arms: SASI bypass group
Procedure: Laparoscopic sleeve gastrectomy — Conventional sleeve gastrectomy using endoscopic stapler
  Arms: Laparoscopic sleeve gastrectomy group

SUMMARY:
Evaluation of the advantages, disadvantages and complications of a recently innovated procedure (Single anastomosis sleeve ileal "SASI" bypass) of the more traditional laparoscopic sleeve gastrectomy "LSG"

DETAILED DESCRIPTION:
Obesity is a major health problem affecting over 1.7 billion people. Obesity is defined as excess body weight due to abnormal or excessive fat accumulation that presents a risk to health. A crude popular measure of obesity is the body mass index (BMI), a person's weight (in kilograms) divided by the square of his or her height (in meters). A person with a BMI of 30 or more is generally considered obese. A person with a BMI equal to or more than 25 is considered overweight.

Obesity is a major risk factor for a number of chronic diseases, including diabetes mellitus, cardiovascular diseases and cancer. It is associated with significant co-morbid conditions and reduced life expectancy. Since 1997, obesity has been officially recognized by the World Health Organization as a global epidemic.

Bariatric surgery has been shown to be the most successful approach in managing morbid obesity that can achieve and sustain great weight loss for a long period.

Common strategies of bariatric surgery are: mechanical obstacles to food ingestion, nutrient-excluded segments and malabsorption, which are a potential cause for complications and should better be avoided from a strictly physiological prospect. Also, such procedures necessitate lifelong medical supervision with the supplementation of vitamins and nutrients. Moreover, they are frequently associated with dysphagia and vomiting as a result of anatomical restrictions.

Laparoscopic sleeve gastrectomy (LSG) was initially established as the first stage of a two stage bariatric approach. It is now used as a primary bariatric procedure because of documented excellent weight loss and an acceptable risk of complication. Advantages include the avoidance of implantable material, maintenance of gastrointestinal continuity, avoidance of malabsorption, and convertibility to other operations. However, The major disadvantage of LSG is the severity of the major postoperative complications like bleeding and staple-line leakage. Staple-line disruption is the most life-threatening complication after LSG, Leaks after sleeve gastrectomy (SG) mostly occur because of the creation of a high internal pressure pouch.

Our understanding of digestive physiology is now changing and the interacting neuroendocrine signals that control hunger, satiety, and energy expenditure are better understood now. The role of GI tract in satiety is a sum of a mechanical sensation of a full stomach, rapidly confirmed by neuroendocrine signals that recognize whether the ingested was indeed nutritive. In terms of meal termination, the most important of these postprandial neuroendocrine signals are an elevation of satiety gut hormones in the blood, such as Glucagon-Like peptide 1 (GLP-1) and Peptide Tyrosine Tyrosine (PYY) and a reduction of ghrelin, an orexigenic hormone mainly produced by neuroendocrine cells mostly located in the gastric fundus. Recent physiological knowledge allows the design of bariatric procedures that aim at neuroendocrine changes instead of mechanical restriction and malabsorption.

"Santoro" have recently reported his long-term data regarding sleeve gastrectomy with transit bipartition (SG þ TB), which is a similar operation to duodenal switch (DS) but without complete exclusion of duodenum in order to minimize nutritional complications. The goal of this operation was to benefit the patients by counterbalancing the harmful effects of the modern diet. Without exclusions and with a simple surgical procedure, SG þ TB amplifies the nutritive stimulation of the distal gut whereas simultaneously diminishing the exposure of the proximal bowel to nutrients without completely deactivating duodenum and jejunum.

A Modification of Santoro's operation was first reported as a case report by Mui in 2013, then as a Case series on 68 patients by Greco and Tacchino in 2014 by performing a loop rather than Roux-en-Y bipartition reconstruction, which came to be known as (Single Anastomosis Sleeve Ileal "SASI") bypass.

That procedure has the advantage of maintaining the natural pathway through the duodenum where a small percentage of food passes, and is associated with minimal post-operative nutritional complications, and allows for full visualization of the biliary system during endoscopy. Moreover, it's suggested that the incidence of leakage and gastroesophageal reflux after sleeve gastrectomy is significantly reduced by the gastroileal bypass due to the decrease in stomach pouch pressure.

This study aims to evaluate SASI bypass as a mode of functional restrictive therapeutic option for morbidly obese patients, versus LSG.

ELIGIBILITY:
Inclusion Criteria:

* Morbid Obesity (BMI ≥ 40 kg/m2) or ( ≥ 35 kg/m2 with associated co-morbidity e.g. type 2 diabetes, joint problems …)
* Age ≥ 18 and < 60
* Failure to achieve adequate and consistent weight loss for at least one year while being followed up by a dietitian.

Exclusion Criteria:

* Patients BMI < 35kg/m2
* Patients who managed to achieve consistent weight loss by diet control.
* Contra-indications to laparoscopic surgery e.g. intolerance to general anesthesia, coagulopathy or an associated condition that requires laparotomy.
* Contra-indications to gastrectomy e.g. gastric ulcer, hiatal hernia or gastro-esophageal reflux disease.
* Previous laparotomy or bariatric procedure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
operative time | the day of operation only
  duration of operation by each technique (in minutes)
intra-operative complications | the day of operation only
  incidence of intra-operative adverse events e.g. bleeding, visceral injury
Post-operative complications | within 12 weeks of the operation
  incidence of post operative complications (Most importantly leakage) other complications e.g. bleeding, thrombo-embolism, chest complications, wound infection...
Percentage of Excess Weight Loss (%EWL) | within 1 year of the operation
  Percentage of weight loss during the year after operation, calculated as a percentage of the excess weight estimated before operation (in kilograms)

SECONDARY OUTCOMES:
change in co-morbidities | within one year of the operation
  defined as when an obesity-related morbidity (e.g. diabetes or dyslipidaemia) becomes resolved after operation, or become controlled with less medication than before operation
incidence of anemia, protein or vitamin deficiency | within one year of the operation
  measured by results of basic lab tests(serum hemoglobin, serum albumin, serum vitamin B12, D, folic acid)

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Elsharkia, Egypt

REFERENCES:
- [Background] Wang Y, Mi J, Shan XY, Wang QJ, Ge KY. Is China facing an obesity epidemic and the consequences? The trends in obesity and chronic disease in China. Int J Obes (Lond). 2007 Jan;31(1):177-88. doi: 10.1038/sj.ijo.0803354. Epub 2006 May 2. PMID 16652128
- [Background] Herron DM. The surgical management of severe obesity. Mt Sinai J Med. 2004 Jan;71(1):63-71. PMID 14770252
- [Background] Santoro S, Milleo FQ, Malzoni CE, Klajner S, Borges PC, Santo MA, Campos FG, Artoni RF. Enterohormonal changes after digestive adaptation: five-year results of a surgical proposal to treat obesity and associated diseases. Obes Surg. 2008 Jan;18(1):17-26. doi: 10.1007/s11695-007-9371-0. Epub 2007 Dec 15. PMID 18080721
- [Background] Brethauer SA, Hammel JP, Schauer PR. Systematic review of sleeve gastrectomy as staging and primary bariatric procedure. Surg Obes Relat Dis. 2009 Jul-Aug;5(4):469-75. doi: 10.1016/j.soard.2009.05.011. Epub 2009 Jun 9. No abstract available. PMID 19632646
- [Background] Fujioka K. Follow-up of nutritional and metabolic problems after bariatric surgery. Diabetes Care. 2005 Feb;28(2):481-4. doi: 10.2337/diacare.28.2.481. PMID 15677821
- [Background] Drazen DL, Woods SC. Peripheral signals in the control of satiety and hunger. Curr Opin Clin Nutr Metab Care. 2003 Nov;6(6):621-9. doi: 10.1097/00075197-200311000-00003. PMID 14557791
- [Background] Casella G, Soricelli E, Rizzello M, Trentino P, Fiocca F, Fantini A, Salvatori FM, Basso N. Nonsurgical treatment of staple line leaks after laparoscopic sleeve gastrectomy. Obes Surg. 2009 Jul;19(7):821-6. doi: 10.1007/s11695-009-9840-8. Epub 2009 Apr 21. PMID 19381737
- [Background] Mui WL, Lee DW, Lam KK. Laparoscopic sleeve gastrectomy with loop bipartition: A novel metabolic operation in treating obese type II diabetes mellitus. Int J Surg Case Rep. 2014;5(2):56-8. doi: 10.1016/j.ijscr.2013.12.002. Epub 2013 Dec 10. PMID 24441436
- [Background] Santoro S, Castro LC, Velhote MC, Malzoni CE, Klajner S, Castro LP, Lacombe A, Santo MA. Sleeve gastrectomy with transit bipartition: a potent intervention for metabolic syndrome and obesity. Ann Surg. 2012 Jul;256(1):104-10. doi: 10.1097/SLA.0b013e31825370c0. PMID 22609843
- [Background] Greco F, Tacchino R. Ileal food diversion: a simple, powerful and easily revisable and reversible single-anastomosis gastric bypass. Obes Surg. 2015 Apr;25(4):680-6. doi: 10.1007/s11695-014-1436-2. PMID 25236398
- See also: Preliminary results from digestive adaptation: a new surgical proposal for treating obesity, based on physiology and evolution — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1516-31802006000400004&tlng=pt
- See also: Bariatric Surgery in Adolescents: Preliminary 1-year Results with a Novel Technique (Santoro III) — https://link.springer.com/article/10.1007%2Fs11695-008-9520-0